CLINICAL TRIAL: NCT01327391
Title: Tolerance of "on Line" Hemodiafiltration and Impact on Morbidity and Cardiovascular Risk Factors in Chronic Renal Failure Patients
Brief Title: Tolerance of "on Line" Hemodiafiltration in Chronic Renal Failure Patients
Acronym: on-line-HDF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UF 7753
Record Dates: First submitted 2008-01-14; First posted 2011-04-01 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2011-03

CONDITIONS: Cardiovascular Disease
Keywords: on line hemodiafiltration; tolerance; quality of life; cardiovascular risk; Hemodialysis patients
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- On line Hemodiafiltration (Active Comparator): Hemodialysis patients treated with on line hemodiafiltration technic
  Interventions: Procedure: On line Hemodiafiltration
- hemodialysis (Other): Hemodialysis patients treated with conventional hemodialysis technic using high flux dialyzers
  Interventions: Procedure: Hemodialysis

INTERVENTIONS:
Procedure: On line Hemodiafiltration — 3 sessions/week; 3-4 hours per session
  Other Names: on line HDF; HDF
  Arms: On line Hemodiafiltration
Procedure: Hemodialysis — 3 sessions/week; 3-4 hours per session; high flux dialyzers
  Other Names: conventional hemodialysis
  Arms: hemodialysis

SUMMARY:
The aim of this study is to appreciate the tolerance of "on line" hemodiafiltration and its impact on morbidity and cardiovascular risk factors in chronic renal failure patient.

DETAILED DESCRIPTION:
The aim of this study is to appreciate the tolerance of "on line" HDF treatment versus conventional high flux hemodialysis in term of adverse events occuring during dialysis sessions between day 30 and day 120 of treatment and to evaluate:

* Quality of life evaluated with the KDQOL questionnaire
* Incidence of cardiovascular events
* Influence of the technic on cardiovascular, inflammatory and infectious risk factors
* Mortality

ELIGIBILITY:
Inclusion Criteria:

* Patient who has signed the written consent form
* Patient aged > 65 and < 90 years
* With creatinine clearance < 10 mL/min
* On dialysis for a minimum of 3 months, with 3 times a week hemodialysis sessions
* Erythropoietin dosage needed to maintain hemoglobin at a constant level (range of hemoglobin: 9-13 g/dL without any variation of more than 2g/dL for less than 3 months)
* Without any problem of vascular access

Exclusion Criteria:

* Patient aged < 65 and > 90 years
* Presence of severe malnutrition (albumin < 20 g/L)
* Unstable clinical condition
* Unipuncture or failed vascular access flow
* Known problems of coagulation

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 415 (Actual)
Dates: Start 2005-05; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
tolerance of "on line" HDF treatment versus conventional high flux hemodialysis in term of adverse events occuring during dialysis sessions | between day 30 and day 120 of treatment

SECONDARY OUTCOMES:
Quality of life evaluated with the KDQOL questionnaire | day 0, 180, 365, 730
Incidence of cardiovascular events | day 180, 365, 730
Influence of the technic on mineral metabolism disturbances | day 180, 365, 730
  measure of mineral metabolism parameters (Ca, PO4, PTH)
All cause and cardiovascular mortality | day 180, 365, 730
Influence of the technic on inflammatory parameters | day 180, 365, 730
  measure of pro-inflammatory cytokines and acute phase reactant proteins
Influence of the technic on microbiological safety | day 180, 365, 730
  measure of microbiological purity of dialysate
Influence of the technic on oxidative stress parameters | day 180, 365, 730
  measure of oxidative stress markers (AOPP, AGE) and antioxidant systems (vitamin E)

CONTACTS AND LOCATIONS:
Overall Officials: Didier AGUILERA, Dr, Study Chair — CHG Vichy France; Lynda AZZOUZ, Dr, Study Chair — CH Roanne France; Jean-Marie BATHO, Dr, Study Chair — CH privé Saint Martin Caen France; Francois COMBARNOUS, Dr, Study Chair — Clinique du Tonkin Villeurbanne France; Lotfi CHALABI, Dr, Study Chair — AIDER Montpellier France; Guy DEGREMONT, Dr, Study Chair — CHG Cambrai France; Maxime HOFFMANN, Dr, Study Chair — Clinique de la Louvière Lille France; Gérard DESCHODT, Dr, Study Chair — AIDER Nimes France; Assia DJEMA, Dr, Study Chair — CHG Cholet France; Alain DUBOUST, Dr, Study Chair — Clinique du Vert Galant, Tremblay en France, France; Alexandre DUMOULIN, Dr, Study Chair — CHLM Beziers France; Baya FADEL-BABBA, Dr, Study Chair — AGDUC La Tronche France; Enrique FIGUEROA, Dr, Study Chair — CH Briancon France; Thierry HAAS, Dr, Study Chair — CMCO Evry France; Jean-Michel HARDIN, Dr, Study Chair — CH Soissons France; Daniel HILLION, Dr, Study Chair — CHI Poissy France; Guillaume JEAN, Dr, Study Chair — CRAT Tassin La Demi Lune France; Véronique JOYEUX, Pr, Study Chair — CHU Pontchaillou Rennes France; Kristian KUNZ, Dr, Study Chair — AURAL France; Antoine LACAILLE, Dr, Study Chair — UNHEP Aulnay sous Bois France; Jacques LEBLEU, Dr, Study Chair — Clinique néphrologique Pont Allant Maubeuge France; Vincent LEMAITRE, Dr, Study Chair — CHG Valenciennes France; Mehadji MAAZ, Dr, Study Chair — CH Louis Pasteur Colmar France; Philippe NICOUD, Dr, Study Chair — Clinique Centre Vallée Blanche Chamonix France; Jean-Paul ORTIZ, Dr, Study Chair — Polyclinique Saint Roch Cabestany France; Jacky POTIER, Dr, Study Chair — CH Louis Pasteur Cherbourg France; Olivier PUYOO, Dr, Study Chair — Clinique Néphrologique Occitanie Muret France; Véronique QUERON, Dr, Study Chair — Polyclinique Francheville Perigueux France; Gilles SCHUTZ, Dr, Study Chair — Centre HD Provence Aubagne France; Francois MAURICE, Dr, Study Chair — CHLM Montpellier France; Bruno SEIGNEURIC, Dr, Study Chair — CHU Larrey Toulouse France; Frederic TOLLIS, Dr, Study Chair — CHU Angers France; Carlos VELA, Dr, Study Chair — CH Perpignan France; Francois WAMBERGUE, Dr, Study Chair — Clinique du Bois Lille France; Christian WOLF, Dr, Study Chair — CH Toulon France; Jean-Paul CRISTOL, Pr, Study Chair — CHU Lapeyronie Montpellier France; Bernard CANAUD, Pr, Principal Investigator — CHU Lapeyronie Montpellier France
Locations (1):
- Centre Hospitalier Universitaire, Montpellier, France